CLINICAL TRIAL: NCT03537300
Title: Efficacy of Deep Cervical Flexor Muscles Training on Neck Pain, Functional Disability and Muscle Endurance in School Teachers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Saud University (Other)
Responsible Party: Principal Investigator, Zaheen A. Iqbal, Principal investigator, King Saud University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RRC-2016-009
Record Dates: First submitted 2018-05-13; First posted 2018-05-25 (Actual); Last update posted 2018-05-25 (Actual); Status verified 2018-05

CONDITIONS: Neck Pain
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental)
  Interventions: Behavioral: DCF muscles training using pressure biofeedback in addition to conventional exercises
- control group (Active Comparator)
  Interventions: Behavioral: conventional exercises

INTERVENTIONS:
Behavioral: DCF muscles training using pressure biofeedback in addition to conventional exercises — DCF muscles training using pressure biofeedback in addition to conventional exercises
  Arms: experimental group
Behavioral: conventional exercises — conventional exercises
  Arms: control group

SUMMARY:
Neck pain (NP) is a common work related disorder. Teaching is one profession in which its prevalence is high. The Daily job of a school teacher involves head down posture while reading, writing, etc., exposing them to risk of developing NP. Deep cervical flexor (DCF) muscles have been shown to have lower endurance in patients with cervical impairment which has been associated with disability. There is limited evidence that reports efficacy of DCF muscles training in occupational NP. This study was done to see the effect of DCF muscles training using pressure biofeedback on pain, muscle endurance and functional disability in school teachers with NP.

DETAILED DESCRIPTION:
Neck pain (NP) is a common work related disorder. Teaching is one profession in which its prevalence is high. The Daily job of a school teacher involves head down posture while reading, writing, etc., exposing them to risk of developing NP. Deep cervical flexor (DCF) muscles have been shown to have lower endurance in patients with cervical impairment which has been associated with disability. There is limited evidence that reports efficacy of DCF muscles training in occupational NP. This study was done to see the effect of DCF muscles training using pressure biofeedback on pain, muscle endurance and functional disability in school teachers with NP. 65 teachers, aged between 25 to 45 years with experience of more than 5 years were agreed to participate in this study. Subjects were randomly divided into two groups, experimental (EG) and control group (CG). In EG, subjects received DCF muscles training using pressure biofeedback in addition to conventional exercises for neck pain while in CG subjects received only conventional exercises. Pain, muscle endurance and disability measured at day 0 (before treatment), day 14 and day 42 after treatment. Endurance of DCF muscles was measured by CCF test using pressure biofeedback instrument, Pain intensity was measured using NPRS and Functional disability was assessed using NDI questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* experience of more than 5 years
* neck pain score of more than 5 on numeric pain rating scale (NPRS), mild to moderate disability score on neck disability index (NDI) and poor cranio-cervical flexion (CCF) test

Exclusion Criteria:

* any neurological sign or symptom, history of spinal surgery or if they were taking any treatment for their pain.

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 65 (Actual)
Dates: Start 2016-05-21 (Actual); Primary Completion 2017-01-01 (Actual); Study Completion 2017-05-01 (Actual)

PRIMARY OUTCOMES:
Change in Pain at day 42, day 14 after intervention from baseline | at day 0 (before treatment), day 14 and day 42 after treatment
  Numeric pain rating scale (NPRS): NPRS. Subjects had to rate their pain on the 0-10 rating scale, where 0 means no pain while 10 is the worst possible pain.
Change in muscle endurance at day 42, day 14 after intervention from baseline | at day 0 (before treatment), day 14 and day 42 after treatment
  Craniocervical flexion test (CCF) test using pressure biofeedback instrument

SECONDARY OUTCOMES:
disability | at day 0 (before treatment), day 14 and day 42 after treatment
  Functional disability was assessed using Neck disability index (NDI) questionnaire. Subjects had to answer the multiple choice questions and their score was interpreted on range from 0 to 50, 0 being no disability and 50 indicating complete disability.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Iqbal ZA, Alghadir AH, Anwer S. Efficacy of Deep Cervical Flexor Muscle Training on Neck Pain, Functional Disability, and Muscle Endurance in School Teachers: A Clinical Trial. Biomed Res Int. 2021 Jan 13;2021:7190808. doi: 10.1155/2021/7190808. eCollection 2021. PMID 33521131